CLINICAL TRIAL: NCT05261243
Title: EEG-characteristics of Neuropsychiatric Symptoms in Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 6/22 S-KH
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Pain
Keywords: Chronic pain; electroencephalography; neuropsychiatry; working memory
MeSH Terms: conditions — Chronic Pain | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EEG / questionnaires / working memory task — EEG resting state measurements and analysis of frequency bands (gamma, beta, alpha, theta), peak frequencies and connectivity measures / questionnaires for depression, anxiety, social activities, cognition, pain, sleep, fatigue / digitalized block-tapping task

SUMMARY:
Chronic pain is a challenge for patients, physicians and society due to its high prevalence and its substantial individual and socio-economic burden.

In recent years, innovative EEG-techniques have been used to study rhythmic brain activities in a variety of neuropsychiatric populations and in chronic pain and various abnormalities in neuronal oscillation patterns and connectivity between brain regions have been observed. However, it remains unclear whether these alterations of brain activity in chronic pain patients reflect pain characteristics like intensity, duration or type (e.g. neuropathic pain), or whether they reflect other symptoms associated with chronic pain.

Neuropsychiatric comorbidities and cognitive deficits of chronic pain are being increasingly recognized, as they frequently cause substantial problems in social life and hinder patients from being able to work. However, it has not been studied yet whether neuronal oscillations and connectivity patterns in the brains of chronic pain patients covary with neuropsychiatric comorbidities (e.g. depression, anxiety, fatigue) and cognitive functioning.

To this end, the investigators will obtain resting state EEG data in large cohort of patients with chronic pain and assess clinical characteristics of chronic pain including a variety of neuropsychiatric symptoms as well as working memory capacity as a proxy for cognitive functioning.

Results from this study will offer valuable insights into and a better understanding of brain dysfunction of patients suffering from chronic pain. This can be helpful for diagnostic and therapeutic advances (e.g. brain stimulation and neurofeedback methods) in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain condition
* Willing and able to sign informed consent for study participation

Exclusion Criteria:

* Severe concomitant neurological or psychiatric disease
* Primary headache condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All chronic pain patients eligible according to the inclusion and exclusion criteria described above treated at the Center for Interdisciplinary Pain Medicine at the Technical University of Munich are invited to voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29 Profile v2.1 (tablet-based) | 1 year (1 assessment per participant)
  29 questions about neuropsychiatric symptoms and quality of life to be rated on a scale from 1-5; higher scores indicate more severe symptoms.
PROMIS-Adult v2.0 - Cognitive Function 4a (tablet-based) | 1 year (1 assessment per participant)
  4 questions about subjective cognitive symptoms to be rated on a scale from 1-5; higher scores indicate more severe symptoms
Working memory task (tablet-based) | 1 year (1 assessment per participant)
  Digitalized self-developed block-tapping task; summarized number of correctly answered levels results in final score (minium 0, maximum 14 points; higher scores indicating higher working memory capacity)
Quantitative resting-state Electroencephalography (5 minute EEG via 29 scalp electrodes): Power Analysis | 1 year (1 assessment per participant)
  Absolute and relative amplitudes/power (gamma, beta, alpha, theta)
Quantitative resting-state Electroencephalography (5 minute EEG via 29 scalp electrodes): Peak Frequency Analysis | 1 year (1 assessment per participant)
  Maximum power value in the EEG frequency spectrum
Quantitative resting-state Electroencephalography (5 minute EEG via 29 scalp electrodes): Connectivity analysis | 1 year (1 assessment per participant)
  Frequency specific connectivity (gamma, beta, alpha, theta)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ploner, Prof. Dr., Principal Investigator — Department of Neurology, Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Department of Neurology, Center for Interdisciplinary Pain Medicine, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will make anonymized data publicly available on data sharing platforms like the Open Science Framework (https://osf.io/)
Supporting Information: Analytic Code
Time Frame: After publication
URL: https://osf.io/

REFERENCES:
- [Background] Ploner M, Sorg C, Gross J. Brain Rhythms of Pain. Trends Cogn Sci. 2017 Feb;21(2):100-110. doi: 10.1016/j.tics.2016.12.001. Epub 2016 Dec 23. PMID 28025007
- [Background] Higgins DM, Martin AM, Baker DG, Vasterling JJ, Risbrough V. The Relationship Between Chronic Pain and Neurocognitive Function: A Systematic Review. Clin J Pain. 2018 Mar;34(3):262-275. doi: 10.1097/AJP.0000000000000536. PMID 28719507
- [Background] Dersh J, Polatin PB, Gatchel RJ. Chronic pain and psychopathology: research findings and theoretical considerations. Psychosom Med. 2002 Sep-Oct;64(5):773-86. doi: 10.1097/01.psy.0000024232.11538.54. PMID 12271108